CLINICAL TRIAL: NCT02627508
Title: Randomized Controlled Pilot Trial of Pregnenolone in Autism
Brief Title: Pilot Trial of Pregnenolone in Autism
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Simons Foundation (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-34762
Record Dates: First submitted 2015-12-02; First posted 2015-12-11 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Autism Spectrum Disorder; Autism; Pregnenolone
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregnenolone (up to 500 mg per day) (Experimental): Twice daily intake of orally administered Pregnenolone will occur on a schedule as described below.
  Weeks 1 and 2: 30mg twice daily (total 60mg per day)
  Weeks 3 and 4: 60mg twice daily (total: 120mg per day)
  Weeks 5 and 6: 90mg twice daily (total: 180mg per day)
  Weeks 7 and 8: 150mg twice daily (total: 300mg per day)
  Weeks 9 and 10: 210mg twice daily (total: 420mg per day)
  Weeks 11 to 14: 250mg twice daily (total: 500mg per day)
  Interventions: Drug: Pregnenolone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — orally administered Pregnenolone capsules
  Arms: Pregnenolone (up to 500 mg per day)
Drug: Placebo — orally administered placebo capsules
  Arms: Placebo

SUMMARY:
This is a research study to examine the tolerability and effectiveness of pregnenolone in individuals with autism. Pregnenolone is a naturally occurring steroid hormone in the brain that has been implicated in treating various psychiatric conditions. The investigators hope to learn the effects and safety of using pregnenolone in reducing irritability and sensitivity to sensory differences and improving social communication in individuals with autism. The investigators hope by studying the effects of pregnenolone in more detail, the investigators can design better ways to treat individuals with autism.

ELIGIBILITY:
Inclusion Criteria:

* outpatients between 14 and 25 years of age with a Tanner stage of IV or V;
* male and female subjects who were physically healthy;
* diagnosis of Autism Spectrum Disorder (ASD) based on DSM-5, expert clinical opinion and confirmed with Autism Diagnostic Interview - Revised (ADI-R) and either Autism Diagnostic Observation Schedule (ADOS) or Childhood Autism Rating Scale (CARS-2);
* Aberrant Behavior Checklist -Irritability (ABC-I)≥ 18 and Clinical Global Impression (CGI)-Severity subscale ≥ 4;
* stable concomitant medications for at least 2 weeks;
* no planned changes in psychosocial interventions during the trial.

Exclusion Criteria:

* Diagnostic and Statistical Manual (DSM-5) diagnosis of schizophrenia, schizoaffective disorder, alcohol use disorder;
* prior adequate trial of pregnenolone;
* active medical problems: unstable seizures (>2 in past month), significant physical illness;
* pregnant or sexually active female subjects who do not adhere to use an appropriate form of external prophylactics;
* participants taking steroid medications.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in parent rated Aberrant Behavior Checklist Irritability (ABC-I) score during treatment | 2-week, 4-week, 6-week, 8-week, 10-week, 14-week

SECONDARY OUTCOMES:
Change from baseline in parent rated Aberrant Behavior Checklist (ABC) scores during treatment | 2-week, 4-week, 6-week, 8-week, 10-week, 14-week
Change from baseline in parent rated Sensory Profile Questionnaire (SPQ) scores during treatment | 2-week, 4-week, 6-week, 8-week, 10-week, 14-week
Change from baseline in Vineland Adaptive Behavior Scales Second Edition (VABS-II) | 2-week, 6-week, 10-week, 14-week
Change from baseline in Clinical Global Impression (CGI) scores during treatment | 2-week, 4-week, 6-week, 8-week, 10-week, 14-week
Change from baseline in levels of pregnenolone and its related neurosteroids in peripheral blood | 14-week
Change from baseline on the Autism Diagnostic Observation Schedule (ADOS) | 14-week
Change from baseline in laboratory based eye-gaze measures | 14-week
Change from baseline in laboratory based electroencephalography (EEG) measures | 14-week
Change from baseline in laboratory clinical lab values including complete metabolic panel, complete blood count with differential, cholesterol panel and routine urinalysis. | 14-week
Change from baseline in parent rated Social Responsiveness Scale (SRS) scores during treatment | 2-week, 6-week, 10-week, 14-week
Change from baseline on the Dosage Record Treatment Emergent Symptom Scale (DOTES) scores during treatment | 2-week, 4-week, 6-week, 8-week, 10-week, 14-week

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes